CLINICAL TRIAL: NCT06636487
Title: Expanding Pulmonary Rehabilitation in Other Chronic Respiratory Disease Than COPD - the ExPuRe Pilot Study
Brief Title: Expand Pulmonary Rehabilitation to Other Chronic Respiratory Diseases Than COPD
Acronym: ExPuRe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Copenhagen University Hospital at Herlev (Other); Amager Hospital (Other); Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Henrik Hansen, Senior Researcher, PhD, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Add-on 96052 to H-22015777
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF); Sarcoidosis; Bronchiectasis; Asthma Bronchiale; Interstitial Lung Diseases (ILD)
Keywords: Pilot RCT Study; Telerehabilitation; home-based pulmonary rehabilitation; pulmonary tele-rehabilitation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Sarcoidosis; Bronchiectasis; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: A randomized clinical, assessor- and statistician blinded multicentre trial with three parallel-groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be informed that the trial is assessing the impact of pulmonary rehabilitation models on predetermined outcomes, but not the specific nature of the models of interest, and the predetermined hypothesis about the purpose, acceptability, willingness and adherence to intervention group allocated.
  All assessors are blinded to group allocation and previous test results. In case of failure keeping the outcome assessor blinded (that is, if a participant reveals his/her allocation) a second assessor will be available to step in and conduct the assessment on another day. To avoid investigators (subconscious) bias the biostatistician who perform the data analyses and validate the results is blinded to group allocation. The research group will interpret the results, before the allocation code is broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pulmonary tele-rehabilitation (PTR) (Experimental): Recieve supervised PTR 2/weekly, session duration of 60 min; 35 min of exercise and 25 min of patient education for 10-weeks. Delivered from Hvidovre/Bispebjerg Hospital to groups of 3 - 5 patients who exercise at home and communicate via tablet-camera. After 10-weeks of PTR, participants are offered once weekly PTR for 60 minutes in groups of 4-8 patients throughout a 65-week maintenance period
  Interventions: Behavioral: pulmonary tele-rehabilitation (PTR)
- Home-based pulmonary rehabilitation (HPR) (Experimental): HPR is an individual self-initiated home-based PR program. Patient goal is to achieve at least 20 min of self-initiated muscle-endurance based exercise 3 days/ weekly for 10-weeks The first session is a home visit by an experienced respiratory physiotherapist and with focus on establishment of exercise goals, formal exercise prescription and education. The home visit is followed by 1/weekly session for 10-weeks.The sessions is delivered from Hvidovre/ Bispebjerg Hospital via tablet-camera or telephone call. After 10-weeks of HPR, participants are offered once weekly PTR for 60 min in groups of 4-8 patients throughout a 65-week maintenance period.
  Interventions: Behavioral: Home-based pulmonary rehabilitation (HPR)
- Control (Active Comparator): Control group will receive usual care; medication, scheduled follow-up visit and possible phone contact with GP or the outpatient respiratory department. Except for assessment visits 10-, 35-, and 75-weeks from baseline no intervention is offered.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: pulmonary tele-rehabilitation (PTR) — PTR is delivered from promoter hospital to a group of 3 - 5 patients who exercise at home and communicate via tablet-camera. Each session is 60 min; 35 min exercise/ 25 min patient education, two times per week for a duration of 10-weeks.
  Specific exercises are evidence-based; been used in several intervention studies on patients with CRD (eg. COPD). Exercises involves larger muscle groups with 50/50 exercises for upper and lower extremities. Volume, intensity and content exercise protocol follow both national and international exercise recommendations. The education sessions consist of dialogue, reflections around empowerment and better living with CRD. Every sixth education session consists of 25 min Mindfulness exercises developed for CRD patients.
  After 10-weeks of PTR, participants are offered once weekly PTR for 60min in groups of 4-8 persons throughout a 65-week maintenance period
  Arms: pulmonary tele-rehabilitation (PTR)
Behavioral: Home-based pulmonary rehabilitation (HPR) — HPR is an individual self-initiated home-based PR aiming to achieve 20 min of self-initiated muscle endurance based exercise; 3-days/weekly for 10-weeks. Exercises are evidence based; used in several intervention studies on patients with CRD (eg. COPD) and involves larger muscle groups with 50/50 exercises for upper/lower extremities.
  First session is a home visit by a respiratory physiotherapist. During the visit the physiotherapist and patient establish exercise goals, exercise prescription and provision of access to mindfulness exercises and an educationbook. The home visit is followed by one weekly session for 10-weeks. A menu of topics relevant to CRD and self-management is discussed. A session is delivered from promoter hospital via tablet-camera or telephone call (patients preference).
  After 10-weeks of HPR, participants are offered once weekly PTR for 60min in groups of 4-8 persons throughout a 65-week maintenance period
  Arms: Home-based pulmonary rehabilitation (HPR)
Behavioral: Control — Receive usual care; medication, scheduled follow up visit and possible phone contact with GP and the outpatient respiratory department. Except for assessment visits 10-, 35-, and 75-weeks from baseline no intervention is offered. If a patient changes their decision and wishes to participate in a conventional hospital- or community-based PR program, it will be granted as this is a highly recommended treatment (e.g. rehabilitation after hospital admitted exacerbation).
  Arms: Control

SUMMARY:
The purpose of this pilot randomized clinical trial is to evaluate the willingness, acceptance, adherence and signs of benefits of structured home-based pulmonary rehabilitation (HPR) and supervised pulmonary tele-rehabilitation (PTR) on respiratory symptoms, quality of life, functioning and physical activity in patients with ILD (Interstitial lung disease, Idiopathic pulmonary fibrosis, Sarcoidosis), Bronchiectasis and Asthma who have a clinically assessed need for a pulmonary rehabilitation program.

The main questions the project aims to answer are:

* Will HPR and PTR appeal to a minimum of 30% of the eligble patients
* Be greatly accepted (≥70% of participant complete 70% or more of the planned sessions) by patients agreeing to participate in the study
* Will PTR and HPR lead to positive changes in respiratory symptom relief, symptom relief in general and improve or maintain physical functioning larger than usual care

Researchers will compare with a comparable control group who gets usual care (scheduled controls and medication but no exercise intervention) to examine the willingness to be randomized and to get an indication on possible health related effects. Participants will be randomly assigned to one of three groups:

1. A structured supervised group-based PTR (exercise twice a week; each session consists of 35 min. evidence-based exercises and 25 min. of patient education)
2. An individual HPR program (self-initiated physical activity) with motivational and professional counseling once a week (10-15min), supported by a tablet screen
3. A control group receiving usual care (CON)

DETAILED DESCRIPTION:
Primary objective of the ExPuRe study is to evaluate the willingness, acceptance, adherence and signs of benefits of structured home-based pulmonary rehabilitation (HPR) and supervised pulmonary tele-rehabilitation (PTR) on respiratory symptoms, quality of life, functioning and physical activity in patients with ILD, Asthma and BE, who have a clinically assessed need for a pulmonary rehabilitation program.

The hypotheses are that HPR and PTR will appeal to 30% of the eligble patients, be greatly accepted (≥70% of participant complete 70% or more of the planned sessions) by patients agreeing to participate in the study, and that PTR and HPR will lead to positive changes in respiratory symptom relief, symptom relief in general and improve or maintain physical functioning larger than usual care, that is the control group (CON - no intervention).

ELIGIBILITY:
Inclusion Criteria:

* Residency in the Capital Region of Copenhagen
* A clinically assessed need for pulmonary rehabilitation including respiratory symptoms, corresponding to MRC grade 2 or higher and where:

  1. Center-based PR is not standard available or
  2. Center-based PR being declined by the patient
* Able to stand up from a chair (height 44-46cm) and walk 10 meters independently (with or without a walking aid)
* Capable of lifting both arms to horizontal with at least 1 kg dumbbells in each hand
* And a minimum of one of the below mentioned diagnoses:

  1. ILD (Interstitial lung disease, Idiopathic pulmonary fibrosis, Sarcoidosis):

     DLCO lower than 80 % or FVC lower than 80%, HRCT verified, Age higher than 40 years, Confirmed respiratory physician diagnosis
  2. Asthma:

     With chronic airway obstruction, ACQ score higher than 1, FEV1 lower than 80%, Age higher than 50 years, Confirmed respiratory physician diagnosis of Asthma
  3. Bronchiectasis:

FEV1 lower than 80%, HRCT verified, Age higher than 40 years, Confirmed respiratory physician diagnosis

Exclusion Criteria:

* Cognitive impairment - unable to follow instructions
* Impaired hearing or vision - unable to see or hear instruction from a tablet
* Unable to understand and speak Danish
* Comorbidities where the exercise content is contraindicated

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Eligibility | Assesment before enrollment
  Number of eligible patients for randomisation (Absolute number)
Adherence | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Number of participants adherent (Participant completion of 70% or more of the planned sessions) (Absolute number)
Acceptability | Acceptance when enrolling the project
  Number of patients accepting to participate (Absolute number)

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) / Chronic Airways Assessment Test (CAAT) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  A patient self administered questionaire. An 8-item questionnaire designed to assess the impact of disease on a person's life (health status). Range of CAT scores from 0-40. Higher scores implicates a more severe impact of COPD on a patient's life(total score point) .
  respiratory symptoms BE (CAT) respiratory symptoms Asthma (CAAT)
Asthma Control Questionnaire (ACQ-7) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  A 7-item asthma specific questionaire to measure the adequacy of asthma control and change in asthma control. Scores range between 0 (totally controlled) and 6 (severely uncontrolled). The ACQ score is calculated as the average of 5, 6 or 7 items (total score point) . Only for those with Asthma
Kings Brief Interstitial Lung Disease | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  The KBILD is a self-completed health status questionnaire that comprises 15 items and a seven-point Likert response scale. It has three domains: psychological, breathlessness and activities and chest symptoms. The KBILD domain and total score ranges are 0-100; 100 represents best health status. (total score point) - only for those with ILD
EuroQol-5D-3L (EQ-5D-3L) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Patient completed questionaires that assess quality of life. Total score from 0-1 on EQ5D- health domain. Total score from 0 - 100 mm on EQ5D-VAS domain. No total domain score.
Multidimensional Fatigue Inventory (MFI-20) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  A patient completed questionaire with a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Items are scored 1-5. In the final score, high scores represent more fatigue (total score point)
Pittsburg Sleep Quality Index (PSQI) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  A self-rated 19-item questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality (total score point).
ActivePAL triaxial accelerometer (PAL) / SENS motion (PAL) (≥50% of total sample | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Wearing time is 24 h per day for 5 days at each time point. Measures sedentary and active body movements, steps per day and METs.
  High number of activity is better
1-minute sit to stand (1-min-STS) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  A clinical test where the patient performes as many sit to stand actions as possible in one minute. Measures endurance by counting the number of repetitions.
30-second sit to stand (30-sec-STS) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  A clinical test where the patient performes as many sit to stand actions as possible in 30 seconds. Measures leg muscle strength by counting the number of repetitions.
Hand-grip strength (Jamar dynamometer) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Measure hangrip muscle strengt in kilo. The higher the better
Number of hospital admissions (respiratory related and all-cause) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Report of the total number
Mortality (respiratory related and all-cause) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Report of the total number
Adverse events | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Report of the numbers of severe adverse events and adverse events
Brief Pain Inventory (BPI) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  A nine item self-administered questionnaire used to evaluate the severity of a patients pain and the impact of this pain on the patients daily functioning. The Every symptom are rated on severity scale ranging from 0 - 10 (total score point).
Short Physical Performance Battery and (SPPB) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  An objective measurement instrument combining three test in one score. The tests consist of a balance test (measured in seconds), lower extremity strength (measured in seconds), and a walkning test measuring functional capacity (measured in seconds) in older adults (65 years of age). Score measured in seconds
Hospital Anxiety and Depression Scale (HADS) | Baseline; At 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Patient self administered questionaires that assess anxiety and depression symptoms. Seven item domain questions for depression with a total score form of 0 - 21 points. Seven item domain questions for anxiety with total score from 0 - 21 points (total score point) .

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Hansen, PhD, Msc, PT, Principal Investigator — Dept. of Respiratory Medicine, University Hospital Hvidovre; Nina Godtfredsen, MD, PhD, Study Chair — Dept. of Respiratory Medicine, University Hospital Hvidovre
Locations (5):
- Denmark (5):
  - Copenhagen University Center, Amager, Copenhagen, Greater Copenhagen
  - Copenhagen University Center, Frederiksberg-Bispebjerg, Copenhagen, Greater Copenhagen
  - Copenhagen University Center, Hvidovre, Copenhagen, Greater Copenhagen
  - Copenhagen University Center, Herlev-Gentofte, Gentofte Municipality, Greater Copenhagen
  - Copenhagen University Center, Hillerød, Hillerød, Greater Copenhagen

IPD SHARING:
Plan to Share IPD: No
Access demands a part application to; (1) Danish Data Protection agency, (2) ethics committee of the capital region, (3) national health Data authorities. Only if the applications are approved data will be considered available for sharing. The investigator will not be able to support this process.